

retonavir tablets and dasabuvir tablets (Viekirax®/Exviera®; Quality of Life measurement using wrist actigraphy in HCV from fatigue and receiving ombitasvir, paritaprevir, and genotype 1 infected, treatment naïve patients suffering 3D regimen): The HEMATITE Study

Statistical Analysis Plan (SAP)

02.05.2018

| Table | Table of Contents |
|-------|------------------------------------------------------|
| Abbre | Abbreviations |
| _ | Introduction3 |
| 2 | Data Sources4 |
| ω | Data Management 4 |
| 3.1 | Handling of Missing Data4 |
| 4 | Objectives4 |
| 4.1 | Primary Objective4 |
| 4.2 | Secondary Objectives4 |
| 5 | Populations 5 |
| 5.1 | Overall Population (OP)5 |
| 5.2 | Analysis Population (AP)5 |
| 6 | Statistical Methods5 |
| 6.1 | Flowchart5 |
| 6.2 | Descriptive Analysis5 |
| 6.3 | Statistical Analysis5 |
| 6.3.1 | Primary Endpoint5 |
| 6.3.2 | Secondary Endpoints5 |
| 6.3.3 | Subgroup Analyses6 |
| 7 | Time table |
| œ | Planned tables and figures for the statistical part7 |

#### **Abbreviations**

| SVR12 | HCV | FSS | EASL | DMP | DB | CRF | BMI | AE | AASLD | 3D regimen |
|---|---|---|---|---|---|---|---|---|---|---|
| Sustained Virologic Response at 12 weeks after end of treatment | Hepatitis C Virus | Fatigue Severity Scale | European Association for the Study of the Liver | Data Management Plan | Database | Case Report Form | Body Mass Index | Adverse event | American Association for the Study of Liver Diseases | Ombitasvir, Paritaprevir, and Ritonavir tablets (Viekirax®); Dasabuvir tablets (Exviera®) |

### 1 Introduction

nervous system (CNS). Data demonstrating a longitudinal change of debilitating physical high priority. This cardinal symptom presents regardless of the stage of liver fibrosis and is to date and are anticipated by the Swiss scientific HCV community. fatigue and increased daytime physical activity upon treatment with 3D regimen are missing hepatic encephalopathy, increasing evidence suggests a direct viral impact on the central difficult to quantify objectively. Similar to other potential reasons for physical fatigue, such as guidelines therefore rate the treatment of HCV patients suffering from debilitating fatigue as a symptom, highly impacting their overall quality of life. AASLD (American Association for the Hepatitis C Virus (HCV) infection reported physical and mental fatigue as the most common Study of Liver Diseases) and EASL (European Association for the Study of the Liver) As described in the HEMATITE study protocol (version V1.0, 09/20/2016) "... patients with

on physical activity of HCV patients suffering from debilitating fatigue. Furthermore, this study manifestations." Switzerland within the next 15 years by creating awareness for patients with extrahepatic supports the Swiss Hepatitis Strategy, which seeks for the elimination of viral hepatitis in The rationale for this observational study is to observe the impact of therapy with 3D regimen

Patients included in this study applied the following criteria:

- Male or female, aged ≥ 18 years
- Treatment-naïve
- Monoinfected with CHCV, GT 1 (confirmed within the last 36 months or at physicians discretion in case of risk factors)
- Non-cirrhotic (based on liver biopsy, fibroscan ≤ 9.6kPa and/or clinical signs)
- . the local Swiss product label prior to any decision to approach the patient to participate in this study. The decision to treat with 3D regimen is made by the physician in accordance with
- Debilitating fatigue (FSS ≥ 4)
- Willing to participate in the study, and willing to wear an activity tracker.

Patients excluded from this study:

- hormonal disorders causing clinically significant fatigue). With sources of fatigue other than HCV (especially, severe depression, cancer and
- investigator's discretion. With conditions that do not allow to adhere to protocol and use of the device at
- Being wheelchair dependent

will be documented in this SAP which will be established and finished by signatures of the Based on the HEMTATITE study protocol details of planned strategies for the data analysis statistician and the principle investigator before data base will be closed

### 2 Data Sources

send to AbbVie Deutschland for electronically data collection in an OpenClinica data base. case report forms (CRFs) for each patient. These CRFs were collected by the monitor and Data sources for the planned analyses are the data documented by the investigators on the

handling of the original data where described in detail in the Data Management Plan (DMP). Physical activity and sleep data will be collected by use of wrist-worn activity trackers transferred in csv format from ActiGraph to the Biostatistik - Tübingen. Dealing with and the activity and (ActiGraph GT9X) which will be processed by device-specific software (ActiLife 6) to obtain sleep-related variables for analysis. These tracker variables will be

### 3 Data Management

## 3.1 Handling of Missing Data

- Missing data from CRFs will be proven within the data collection in OpenClinica and clarified by queries to the monitoring.
- less than two eligible weeks are available, daytimes variables of previous weeks will For tracker variables datasets of two eligible weeks (10 working days) are needed. If be used.
- No other replacement of missing data will take place

### 4 Objectives

### 4.1 Primary Objective

According to the HEMATITE study protocol (version V1.0, 09/20/2016) the primary objective regimen between baseline (before treatment start) and post-treatment week 12". is "to observe changes in physical activity in patients with newly initiated therapy with 3D

## 4.2 Secondary Objectives

The secondary objectives include the following endpoints:

- To correlate subjective fatigue (assessed by means of FSS) and physical activity of treatment with 3D regimen. (measured with an electronic activity tracker) at baseline, during and after 12 weeks
- after treatment with 3D regimen (defined as HCV not detectable, 12 weeks after the To observe the proportion of patients achieving sustained virologic response (SVR12) last dose of 3D regimen).
- during and after 12 weeks of treatment with 3D regimen To observe sleep efficiency (assessed by means of activity tracker) at baseline,

### 5 Populations

## 5.1 Overall Population (OP)

analyzed for this population. meeting all inclusion and no exclusion criteria. Descriptive and safety parameters will be The overall population consists of all documented patients signing the informed consent and

# 5.2 Analysis Populations (ITT and mITT)

overall population with treatment as intended to protocol and received study medication at modified ITT population (mITT) as well. The ITT consists of all documented patients of the secondary endpoints will be analyzed for mITT. visits. For ITT and mITT descriptive and safety parameters will be analyzed. Primary and least once. Additionally, mITT consists of all patients of the ITT which take part at all five The statistical analyses will be performed for the intention-to-treat population (ITT) and the

### Statistical Methods

### 6.1 Flowchart

The formation of the populations will be described by a Consort-Flowchart.

## 6.2 Descriptive Analysis

missings (miss), total and relative frequency. median and q3). Qualitative parameters will be presented with number (N), number of missings (miss), mean, standard deviation, minimum, maximum and quartiles (q1, q2 = The results of descriptive analyses will be shown in common tables for the populations OP, and mITT where quantitative parameters will be shown with number (N), number of

## 6.3 Statistical Analysis

### 6.3.1 Primary Endpoint

level will be set to  $\alpha = 0.05$ , the test will be performed two-sided. or Wilcoxon-test, depending from the distribution of the data (normal or not). The significance (before treatment start) and post-treatment week 12, will be calculated and analyzed by t-test The primary endpoint, the change of the mean daytime physical activity between baseline

## 6.3.2 Secondary Endpoints

the difference between baseline and the respective follow-up visits will be calculated and For the secondary endpoints "change of FSS between baseline, during and after 12 weeks"

parameters daytime activity and sleep efficiency. shown with 95% confidence intervals (95%-CI). This analysis will also be performed for the

baseline, during the study and after 12 weeks. Furthermore for daytime activity, FSS and sleep efficiency 95%-Cl will be provided at

correlation coefficient visit and for the changes between baseline and follow-up visits using Spearman's rank The correlation between mean daytime physical activity and FSS will be analyzed for each

confidence interval. The proportion of patients achieving SVR12 will be calculated and shown with 95

## 6.3.3 Subgroup Analyses

regimen". These analyses will be performed for ITT and mITT. According to the HEMATITE study protocol (version 1.0, 09/20/2016) "subgroup analyses will provided for patients who achieve/do not achieve SVR12 after treatment with 3D

Daytime activity, FSS and sleep efficiency will be compared between following groups

- Patients with Ribavirin vs. patients without Ribavirin at visit V2, V3, V4 and V5
- Women vs. men at each visit.
- Patients with different fibrosis stages (F0, F1, F2 or F3) at each visit
- Patients with different age categories (median split) at each visit

Additionally for patients with GT1a vs. patients with GT1b FSS will be compared at each visit.

All statistical analyses will be performed by SPSS® for Windows, version 22.0

### 7 Time table

The following temporary periods of time are planned:

| Integrated Clinical Study Report | Statistical analyses | Cleanfile | Data input until | Last patient out |
|---|---|---|---|---|
| September 2018 | Juli/August 2018 | June 2018 | May 2018 | April 2018 |

Deviations from this plan because of unexpected occurence are possible

# 8 Planned tables for the statistical part

| Number | r Items | Database/Variables |
|---|---|---|
| 1 Info | Information to the study course | |
| 1.1 | Enrolled/dropped out patients | Database 1 – Visit 1 (Day -28) |
| 1.2 | Study visits and study termination | Database 1 - Visit 1 (Day -28) - Visit 5 |
| 3 | | R12) |
| C | ratient eligibility criteria | Database 1 – visit 1 (Day -28) |
| | atterns baseline characteristics | |
| 2.1 | Demographics | Database 1 – Visit 1 (Day -28) |
| 2.2 | Medical history | Database 1 – Visit 1 (Day -28) |
| 2.3 | Fatigue severity scale (FSS) | Database 1 – Visit 1 (Day -28) |
| 2.4 | HCV history | Database 1 – Visit 1 (Day -28) |
| 2.5 | Vital signs | Database 1 – Visit 1 (Day -28) |
| 2.6 | Laboratory | Database 1 – Visit 1 (Day -28) |
| 2.7 | Smoking/alcohol status | Database 1 – Visit 1 (Day -28) |
| 2.8 | Activity tracker | Database 2 – Tracker data |
| 2.9 | Concomitant medication | Database 1 – Visit 1 (Day -28) |
| 3 Patio | Patients characteristics during study | |
| 3.1 | Activity tracker | Database 2 – Tracker data |
| 3.2 | (S)AEs and concomitant medication | Database 1 – Visit 2 (Day 1) – Visit 5 (Day 168, SVR12) |
| 3.3 | Fatigue severity scale (FSS) | Database 1 – Visit 2 (Day 1) – Visit 5 (Day 168, SVR12) |
| 3.4 | Start of 3D regimen / 3D regimen | Database 1 – Visit 2 (Day 1) – Visit 4 (Day 84) |
| 3.5 | Vital signs | Database 1 - Visit 2 (Day 1) - Visit 5 (Day 168, SVR12) |
| 3.6 | Laboratory | Database 1 - Visit 2 (Day 1) - Visit 5 (Day 168, SVR12) |
| 3.7 | Physical examination | Database 1 – Visit 4 (Day 84) and Visit 5 (Day 168, SVR12) |
| 3.8 | Smoking/alcohol status | Database 1 – Visit 5 (Day 168, SVR12) |
| 4 Stati | Statistical analysis | |
| 4.1 | Primary endpoint | Database 2 - Tracker data |
| 4.2 | Secondary endpoints – Change of parameters | Database 1 (visit data) and database 2 (tracker data) |
| 4.3 | Secondary endpoints - Correlations | Database 1 and database 2 |
| 4.4 | Secondary endpoints - Proportion of SVR12 | - |

| Number Items | Items | Database/Variables |
|---|---|---|
| 5 Subgi | 5 Subgroup analyses | |
| 5.1 | Daytime activity, FSS and sleep efficiency for patients with/without Ribavirin | Database 1 and database 2 |
| 5.2 | Daytime activity, FSS and sleep efficiency for Women vs. men | Database 1 and database 2 |
| 5.3 | Daytime activity, FSS and sleep efficiency for patients with different fibrosis stages | Database 1 and database 2 |
| 5.4 | Daytime activity, FSS and sleep efficiency for patients with different age categories | Database 1 and database 2 |
| 5.5 | FSS for patients with GT1a vs. GT1b | Database 1 and database 2 |